CLINICAL TRIAL: NCT00827736
Title: Botulin Toxin Versus Isosorbidedinitrate Ointment in Treatment Anal Fissure; A Prospective, Blinded, Randomized Trial
Brief Title: Comparison of Treatment Success of Botox Injection in the Internal Sphincter Versus Isosorbidedinitrate Ointment in Patients With an Anal Fissure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouwe Gasthuis (Other)
Responsible Party: S.Festen, MD, Onze Lieve Vrouwe Gasthuis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00.058
Record Dates: First submitted 2009-01-20; First posted 2009-01-23 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Anal Fissure
Keywords: anal fissure; fissura ani; botox; ISDN; Nitric oxide donor
MeSH Terms: conditions — Fissure in Ano | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox injection (Experimental): injection of 10U of BT (Botox®; Allergan, Irvine, California, USA) in the IAS on each side of the anterior midline. In addition, a placebo ointment has to be applied to the anoderm six times a day
  Interventions: Procedure: Botox
- ISDN ointment (Active Comparator): application of ISDN 1% ointment 6 times a day. injection of placebo into internal anal sphincter
  Interventions: Procedure: Botox; Drug: ISDN ointment; Drug: Placebo

INTERVENTIONS:
Procedure: Botox — injection of 10U of BT (Botox®; Allergan, Irvine, California, USA) in the IAS on each side of the anterior midline.
Drug: ISDN ointment — application of ISDN 1% ointment 6 times a day
  Arms: ISDN ointment
Drug: Placebo — Injection of placebo into internal anal sphincter (ISDN ointment arm)
  Applied to the anoderm six times a day (Botox injection arm)
  Arms: ISDN ointment

SUMMARY:
The standard treatment of anal fissure in the netherlands (ISDN ointment) is being compared to a relatively new treatment (injection of Botox in the internal anal sphincter). The study hypothesis is that after 4 months, Botox has healed more patients than ISDN. The comparison is done blinded for the surgeon and the patient.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients over the age of 18 with a chronic anal fissure presenting to our surgical outpatient clinic

Exclusion Criteria:

* pregnancy
* previous anal surgery
* Crohn's disease
* systemic causes of an anal fissure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2002-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
macroscopic healing of the fissure | 4 months

SECONDARY OUTCOMES:
complications | 12 months
fissure recurrence | 12 months
fissure related pain | 12 months
costs | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael Gerhards, MD, Study Director — Onze Lieve Vrouwe Gasthuis
Locations (1):
- Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Result] Brisinda G, Maria G, Bentivoglio AR, Cassetta E, Gui D, Albanese A. A comparison of injections of botulinum toxin and topical nitroglycerin ointment for the treatment of chronic anal fissure. N Engl J Med. 1999 Jul 8;341(2):65-9. doi: 10.1056/NEJM199907083410201. PMID 10395629